CLINICAL TRIAL: NCT00002064
Title: Toxoplasmic Encephalitis in Patients With AIDS. Treatment and Prevention of Relapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Medical Foundation (Other)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 021A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1989-06

CONDITIONS: Toxoplasmosis, Cerebral; HIV Infections
Keywords: Sulfonamides; Toxoplasmosis; AIDS-Related Opportunistic Infections; Pyrimethamine; Drug Therapy, Combination; Encephalitis; Acquired Immunodeficiency Syndrome; Clindamycin
MeSH Terms: conditions — Toxoplasmosis, Cerebral; HIV Infections; Toxoplasmosis; AIDS-Related Opportunistic Infections; Encephalitis; Acquired Immunodeficiency Syndrome | interventions — Pyrimethamine; Clindamycin

INTERVENTIONS:
Drug: Pyrimethamine
Drug: Clindamycin

SUMMARY:
To compare pyrimethamine and intravenous (IV) clindamycin vs. pyrimethamine and sulfonamides in the treatment of AIDS patients with central nervous system (CNS) Toxoplasma gondii.

ELIGIBILITY:
Exclusion Criteria

Co-existing Condition:

Patients with the following conditions are excluded:

* Opportunistic infection (Pneumocystis carinii pneumonia (PCP), cryptococcal meningitis) or other conditions (brain abscess) which would make treatment results difficult to interpret due to concurrent infection, disease, or therapy.

Patients with other opportunistic infections or brain diseases are excluded.

Patients with AIDS and cerebral toxoplasmosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Palo Alto Med Foundation, Palo Alto, California, United States